CLINICAL TRIAL: NCT01806116
Title: Decitabine for Myelodysplastic Syndromes and Acute Myeloid Leukemia Before Allogeneic Hematopoietic Cell Transplantation
Acronym: DFMBHSCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hematology-01
Record Dates: First submitted 2013-03-05; First posted 2013-03-07 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Higher-risk Myelodysplastic Syndrome; Relapsed /Refractory Acute Myeloid Leukemia
Keywords: myelodysplastic syndrome; higher-risk; acute myeloid leukemia; relapsed /refractory; decitabine; hematopoietic cell transplantation; bridge therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Decitabine

ARMS (1):
- decitabine + transplantation (Experimental)
  Interventions: Drug: decitabine

INTERVENTIONS:
Drug: decitabine

SUMMARY:
Allogeneic stem cell transplantation (SCT) is the only potentially curative therapy for patients with myelodysplastic syndrome (MDS) and acute myeloblastic leukemia (AML). Relapse remains a leading cause for treatment failure after hematopoietic cell transplantation (HCT) in patients，so that there is the need to continue to look for alternative therapies. Decitabine, is known to inhibit DNA methyltransferase which results in DNA hypomethylation and expression of silenced genes including those involved in apoptosis. The approval of decitabine for the treatment of MDS and AML has provided an alternative strategy to inhibit disease progression in transplant-eligible patients. To assess the effect of pretransplant decitabine treatment on post transplant outcomes, we recently reviewed our institutional experience with MDS and AML patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 8- 65 years
* Diseases must be myelodysplastic syndrome and acute myelocytic leukemia
* Must need a bone marrow transplant
* Must have the ability to observe the efficacy and events
* Patient must have ability to understand and willingness to provide written informed consent prior to participation in the study and any related procedures being performed

Exclusion Criteria:

* Must not have uncontrolled intercurrent illness including ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements
* Must not be pregnant or breastfeeding; pregnant women are excluded from this study because decitabine is a Category D agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with decitabine, breastfeeding should be discontinued if the mother is treated with decitabine; these potential risks may also apply to other agents used in this study
* Must not have a known or suspected hypersensitivity to decitabine

Ages: 8 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-09; Primary Completion 2013-03 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
overall survival rates | three years

SECONDARY OUTCOMES:
disease free survival | three years

OTHER OUTCOMES:
The incidences of acute and chronic graft-versus-host disease | three years

CONTACTS AND LOCATIONS:
Overall Officials: Wu depei, Phd, Principal Investigator — First Affiliated Hospital, Soochow University